CLINICAL TRIAL: NCT06002737
Title: The Safety and Effectiveness of Using Ultrasound Scalpel to Coagulate 5-7mm Blood Vessels : a Prospective, Multicenter Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hecheng Li M.D., Ph.D (Other)
Collaborators: Ruijin Hospital (Other); Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other); Zhejiang University (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor-Investigator, Hecheng Li M.D., Ph.D, Prof, Ruijin Hospital
Organization: Ruijin Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTS-018
Record Dates: First submitted 2023-08-16; First posted 2023-08-21 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: The Safety of Ultrasound Knife Coagulation for Blood Vessels With a Diameter Greater Than 5mm and Less Than or Equal to 7mm

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Arm 1 (Experimental): Using Experimental harmonic scalpel to dissect the vessel
  Interventions: Device: Occlusion of blood vessels with a diameter greater than 5mm and less than or equal to 7mm using harmonic scalpel
- Arm 2 (Active Comparator): Using Harmonic Ace+7(Ethicon Endo-Surgery, LL), 5mm Diameter Shears with Advanced Hemostasis to dissect the vessel
  Interventions: Device: Occlusion of blood vessels with a diameter greater than 5mm and less than or equal to 7mm using harmonic scalpel

INTERVENTIONS:
Device: Occlusion of blood vessels with a diameter greater than 5mm and less than or equal to 7mm using harmonic scalpel — Screening of lung or esophageal surgery patients who meet the inclusion criteria but do not meet the exclusion criteria, and evaluating the effectiveness and safety of ultrasound scalpel in the process of coagulation of blood vessels with a diameter greater than 5mm but not equal to 7mm.

SUMMARY:
Evaluation of the safety and effectiveness of disposable ultrasound soft tissue cutting and hemostasis equipment for coagulating 5-7mm blood vessels with ultrasound scalpel tips

DETAILED DESCRIPTION:
Screening lung and esophageal surgery patients who must meet the inclusion/exclusion criteria, and evaluating the effectiveness and safety of ultrasound scalpel in the process of 5-7mm blood vessel disconnection and occlusion

ELIGIBILITY:
Inclusion Criteria:

* 1) 18 years old ≤ age ≤ 75 years old, regardless of gender;

  2) Based on the preoperative CT examination results, it is determined that the patient has at least one blood vessel that needs to be coagulated during the surgery, with a diameter greater than 5mm but less than or equal to 7mm;

  3) Before the start of the study, the patient is willing and able to sign an informed consent form approved by the ethics committee;

  4) The patient understands the clinical study, cooperates with the research procedure, and is willing to conduct postoperative follow-up according to the protocol.

Exclusion Criteria:

* 1) Patient body mass index (BMI) ≥ 35.0 kg/m2;

  2) Prothrombin time greater than 5 seconds;

  3) Researchers have determined that the tumor may invade the target blood vessel, which may affect the operation or effectiveness of vascular occlusion and disconnection;

  4) Researchers have determined that there may be variations, deformities, or calcifications in the target vessel that may affect the evaluation of the primary endpoint, which may affect the operation or effectiveness of vascular occlusion and disconnection;

  5) Patients receive preoperative chemotherapy and radiation therapy;

  6) Patient's fasting blood glucose ≥ 11.1mmol/l;

  7) Hypertensive patients' blood pressure has not been effectively controlled, and their blood pressure is ≥ 140/90 millimeter of mercury （mmHg） in a stable state after medication;

  8) Pregnant or lactating women, or women with pregnancy plans during the trial period;

  9) Participated in other clinical studies within 3 months;

  10) Individuals with mental disorders and lack of autonomous behavioral ability;

  11) Other researchers believe that it is not suitable to participate in the experiment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2024-04-18 (Actual)

PRIMARY OUTCOMES:
The success rate of successful coagulation and disconnection of target blood vessels using ultrasound knife | From the target Vascular detachment to finish of the surgery
  The success rate is defined as the number of subjects who successfully occluded and severed blood vessels divided by the number of subjects in the analysis dataset. Each subject should use an ultrasound knife to occlude and sever at least one target vessel

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Jiao Tong University School of Medicine Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li C, Niu Z, Xu J, Yao J, Yan Y, Chang Z, Wang X, Jing H, Han D, Zhang Y, Che J, Lin J, Wang M, Fan J, Hu J, Li H. Evaluation of ultrasonic energy for sealing 5-7 mm blood vessels in thoracoscopic surgery: a noninferiority randomized controlled trial. Transl Lung Cancer Res. 2025 Sep 30;14(9):3636-3644. doi: 10.21037/tlcr-2025-433. Epub 2025 Sep 25. PMID 41133002
- [Derived] Wang X, Li C, Fan J, Hu J, Wang M, Li H. Safety and effectiveness of using Disposable Ultrasonic shears to coagulate 5-7 mm blood vessels: protocol for a prospective, multicenter, randomized, parallel controlled, non-inferiority clinical trial. BMC Surg. 2024 Jul 19;24(1):212. doi: 10.1186/s12893-024-02497-x. PMID 39030560